CLINICAL TRIAL: NCT06760923
Title: Urinary Proteomic Assessment of Ovarian Malignancy and Disease Progression
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024040383
Record Dates: First submitted 2024-12-27; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Ovarian Cancer (OvCa)
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnosis undetermined: Patients who are initially diagnosed with conditions such as "pelvic mass" or "malignant ascites," which may suggest ovarian cancer, or those who are initially diagnosed with conditions such as "ovarian cyst," "hydrosalpinx," "uterine fibroids," or "adenomyosis," which are considered non-malignant gynecological diseases, and who have not yet undergone any surgery or treatment.

SUMMARY:
The goal of this observational study is to determine the urinary proteomic characteristics in women with and without ovarian cancer. The main questions it aims to answer are:

1. What is the difference in urinary protein composition between patients with ovarian cancer and those without it?
2. Can these differences in urinary protein composition aid in the diagnosis of ovarian cancer?
3. Are urinary protein markers associated with tumor burden in urine samples from patients with ovarian cancer?
4. Can urinary protein markers be used for disease surveillance in ovarian cancer patients?

ELIGIBILITY:
Inclusion Criteria:

* Female patients in the gynecological ward for surgical treatment.
* Initial diagnosis of "pelvic mass" or "malignant ascites" may be considered as ovarian cancer; Or the initial diagnosis of "ovarian cyst", "hydrosalpinx", "uterine fibroids" or "uterine adenomyosis" are considered as gynecological non-malignant diseases.
* Over 18 years of age.
* Voluntary participation and signing of informed consent.

Exclusion Criteria:

* Study participants with a prior history of malignant tumors.
* Study participants with prior chronic kidney disease or renal insufficiency.
* Study participants who have received or are receiving treatment for primary disease.
* Study participants whose pathological diagnosis was not clear.

Any patient should be excluded from the study if:

* Study participants withdraw informed consent and request withdrawal.
* Study participants were unable to provide a qualified urine sample.
* There are situations in which the researcher considers it necessary to withdraw from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological diagnosis | From enrollment to the end of surgery or biopsy at 1 weeks
  The histological type of the disease is confirmed by surgery or biopsy

SECONDARY OUTCOMES:
Progression | From enrollment to the end of treatment at 6 months
  Patients with ovarian cancer who have recurrent disease after initial treatment with serological or imaging evidence

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hosipital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
The affiliation has not approved to share individual participant data